CLINICAL TRIAL: NCT05830578
Title: Clinical Validation of the Electrocardiogram Measurement and Atrial Fibrillation Detection Function of a Wearable Smartwatch
Brief Title: Clinical Validation of the Electrocardiogram Measurement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ECG and AF Validation
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation
Keywords: Electrocardiogram; Atrial Fibrillation; Validation; Software as Medical Device (SaMD)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Subjects enrolled into Cohort 1 must have no known medical history of AFib and in normal sinus rhythm at the time of screening.
  Interventions: Device: ASUS Blood Pressure Monitor/Oximeter/ECG Monitor
- Cohort 2: Subjects enrolled into Cohort 2 must have a known diagnosis of persistent or permanent AFib and be in AFib at the time of screening.
  Interventions: Device: ASUS Blood Pressure Monitor/Oximeter/ECG Monitor

INTERVENTIONS:
Device: ASUS Blood Pressure Monitor/Oximeter/ECG Monitor — The ASUS Blood Pressure Monitor/Oximeter/ECG Monitor analyzes data collected by the integrated electrical sensors on a ASUS Vivowatch to generate an ECG waveform similar to a Lead I, calculate average heart rate, and provide a rhythm classification to the user for a given 30 second session. When a user opens the ECG App while wearing the ASUS VivoWatch on one wrist and places the finger of the opposite hand on the digital crown, they are completing the circuit across the heart which begins a recording session.
  Once the recording session is complete, the ECG App performs signal processing, feature extraction and rhythm classification to generate a session result.

SUMMARY:
Atrial fibrillation (AFib) is a common type of cardiac arrhythmia in clinical practice, affecting millions of people worldwide. Early detection and treatment of atrial fibrillation are crucial in preventing serious complications such as stroke and heart failure. In recent years, with the flourishing development of wearable devices and mobile technology, electrocardiogram (ECG) measurement applications embedded in smartwatches have gradually become a non-invasive and convenient method for heart rate monitoring. However, the accuracy of these devices has not yet been fully determined. This study aims to verify the ECG measurement and atrial fibrillation detection function of the ASUS Blood Pressure Monitor/Oximeter/ECG Monitor. The accuracy of the ECG application in detecting atrial fibrillation and measuring ECG will be evaluated by comparison with standard 12-lead ECGs.

DETAILED DESCRIPTION:
This study plans to recruit 602 adults over the age of 22. All participants will undergo heart rate measurements using both the smartwatch ECG application and the 12-lead ECG. The heart rate measurement using the ECG application will be operated by the participants themselves under the guidance of the testing personnel. The 12-lead ECG will be operated by trained medical professionals. The results of the heart rate measurement from both devices will be recorded synchronously, and the consistency of heart rate interpretation and ECG waveforms between the smartwatch ECG application and the 12-lead ECG measurement will be compared to verify the accuracy of the ECG application.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to participate in the study procedures as described in the consent form
* Individuals who are 22 years of age and older at time of screening
* Able to communicate effectively with and follow instructions from the study staff
* Subjects enrolled into Cohort 1 must have no known medical history of AFib and in normal sinus rhythm at the time of screening.
* Subjects enrolled into Cohort 2 must have a known diagnosis of persistent or permanent AFib and be in AFib at the time of screening.

Exclusion Criteria:

* Physical disability that precludes safe and adequate testing
* Mental impairment as determined by the Investigator
* Pregnant women at the time of the screening visit.
* Subjects with any Medical History, Physical exam, vital sign or any other study procedure finding/assessment that in the opinion of the investigator could compromise subject safety during study participation or interfere with the study integrity and/or the accurate assessment of the study objectives. This includes patients with known untreated medical conditions that are considered clinically significant by the Investigator, such as but not limited to significant anemia, important electrolyte imbalance and untreated or uncontrolled thyroid disease. Physical exam limitations include but not limited to open wound(s) on the wrist and forearm where the subject will be wearing the watch.
* Any history of wrist surgery with scarring in the area of the sensor location on the wrist where the subject will be wearing the watch.
* Vital signs measurement, medical history, or physical exam finding that makes the subject inappropriate for participation according to the Investigator.
* Tattoos or moles in the area of the sensor location on the wrist where the subject will be wearing the watch.
* Skin conditions on either wrist that would preclude subject from wearing watch on either wrist. Severe symptomatic (or active) overly dry/injured skin, skin disorders, or allergic skin reactions such as eczema, rosacea, impetigo, dermatomyositis or allergic contact dermatitis on wrist and locations where the electrodes will be placed (e.g. chest, forearms, stomach), as determined by the investigator.
* Known allergy or significant sensitivity to medical adhesives, isopropyl alcohol, or ECG patch.
* Clinically significant hand tremors as judged by the Investigator.
* Subjects with implanted cardiac devices such as a Pacemaker or an automated Implantable Cardioverter - Defibrillator.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include two cohorts of subjects:
  1. Cohort 1 will include subjects with no known history of AFib and are in normal sinusn rhythm at time of screening.
  2. Cohort 2 will include subjects with known persistent or permanent or chronic AFib who are in AFib at the time of screening.
  The study will enroll equal subjects with and without a known diagnoiss of AFib into two separate cohorts. A total of 602 subjects will be recruited (301 for SR cohort and 301 for AFib cohort).
  The following age and gender enrollment targets will be adhered to during subject recruitment:
  1. A minimum of 20% of subjects in both cohorts will be enrolled in each of the age categories of 55 to 64, and ≥65 years, and a minimum of 10% of subjects in both cohorts in the age category of <55 years.
  2. At least 40% of subjects in Cohort 1 will be female. At least 20% of subjects in Cohort 2 will be female.
Sampling Method: Non-Probability Sample
Enrollment: 602 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the ECG App algorithm | One day visit
  Sensitivity and specificity of the ECG App algorithm in detecting AFib compared with physician-adjudicated 12-lead ECG will be calculated.

IPD SHARING:
Plan to Share IPD: No